CLINICAL TRIAL: NCT03025165
Title: A Comparison of Different Community Models of ART Delivery Amongst Stable HIV+ Patients in Two Urban Settings in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPTN 071c
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community Adherence Clubs (Experimental): ART adherence support, symptom screening and dispensation of pre-packed medications by community health worker to a club meeting of 20-25 HIV+ patients every three months, with two clinic visits every year for clinical review and laboratory monitoring
  Interventions: Other: Community Adherence Clubs
- Home-Based ART Delivery (Experimental): Individuals receive ART adherence support, symptom screening and dispensation of pre-packed medications by community health worker at their household every three months, with two clinic visits every year for clinical review and laboratory monitoring
  Interventions: Other: Home-Based ART Delivery
- Standard of Care (Other): Delivery of ART adherence support, symptom screening and dispensation of medications at the local clinic according to local guidelines.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Community Adherence Clubs — Provision of ART care in the community to a club of 20-25 HIV+ patients
  Arms: Community Adherence Clubs
Other: Home-Based ART Delivery — Provision of ART care to an individual at their home
  Arms: Home-Based ART Delivery
Other: Standard of Care — Delivery of ART adherence support, symptom screening and dispensation of medications at the local clinic according to local guidelines.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to compare the virological and clinical outcomes of patients participating in community models of ART delivery to the standard of care in an urban setting in Zambia.

DETAILED DESCRIPTION:
The outcomes of this study will be measured in a prospective cohort of adult patients enrolled into ART care in two urban communities participating in the HPTN 071 (PopART) trial. The two community models are: 1) adherence clubs, groups of 20-25 stable patients who receive ART care in the community every 3 months, and 2) home-based ART delivery in which a community health worker delivers ART care to an individual at home every 3 months. The standard of care is delivery of ART care at the local clinic.

ELIGIBILITY:
Inclusion Criteria:

18 years or older On first-line ART and retained in care for more than 6 months Virologically suppressed World Health Organization (WHO) stage I and II at time of screening Reside within the clinic catchment area Willing to provide written informed consent and accept Community HIV-care Provider (CHiPs) intervention

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2526 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | One year after beginning participation in the program
  Viral suppression at 12 months measured using the standard of care viral load testing equipment currently in place. Viral suppression will be defined according to National guidelines.

SECONDARY OUTCOMES:
Viral suppression at 24 months | Two years after beginning participation in the program
  Undetectable HIV viral load 24 months after entry into the models of care. This will be done as part of routine laboratory monitoring and measured using routine programmatic data.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Limbada, MBCHB, MScID, Principal Investigator — Zambart
Locations (1):
- Zambart, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Limbada M, Macleod D, Situmbeko V, Muhau E, Shibwela O, Chiti B, Floyd S, Schaap AJ, Hayes R, Fidler S, Ayles H; HPTN 071 (PopART) study team. Rates of viral suppression in a cohort of people with stable HIV from two community models of ART delivery versus facility-based HIV care in Lusaka, Zambia: a cluster-randomised, non-inferiority trial nested in the HPTN 071 (PopART) trial. Lancet HIV. 2022 Jan;9(1):e13-e23. doi: 10.1016/S2352-3018(21)00242-3. Epub 2021 Nov 26. PMID 34843674
- [Derived] Limbada M, Bwalya C, Macleod D, Floyd S, Schaap A, Situmbeko V, Hayes R, Fidler S, Ayles H; HPTN 071 (PopART) Study Team. A comparison of different community models of antiretroviral therapy delivery with the standard of care among stable HIV+ patients: rationale and design of a non-inferiority cluster randomized trial, nested in the HPTN 071 (PopART) study. Trials. 2021 Jan 12;22(1):52. doi: 10.1186/s13063-020-05010-w. PMID 33430928

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03025165/Prot_ICF_000.pdf